CLINICAL TRIAL: NCT02902497
Title: Impact of the Surgical Experience on Cochleostomy Location: A Comparative Temporal Bone Study Between Endaural and Posterior Tympanotomy Approaches for Cochlear Implantation
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 15-METHODO-01
Record Dates: First submitted 2016-08-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Cochlear Implantation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study was to evaluate, in the hands of an inexperienced surgeon, the cochleostomy location of an endaural approach (MINV) compared to the conventional posterior tympanotomy (MPT) approach. Since 2010, the investigators use in the ENT department of Nice a new surgical endaural approach to perform cochlear implantation. In the hands of an inexperienced surgeon, the position of the cochleostomy has not yet been studied in detail for this technique. This is a prospective study of 24 human heads. Straight electrode arrays were implanted by an inexperienced surgeon: on one side using MPT and on the other side using MINV.

ELIGIBILITY:
Inclusion Criteria:

* cadaver heads
* person had provided written consent to give their entire body to science

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cadaver heads
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
position of the cochleostomy | at 1 day

IPD SHARING:
Plan to Share IPD: No